CLINICAL TRIAL: NCT00868855
Title: The Intracoronary Tissue-type Plasminogen Activator (t-PA) Release Predicts Major Adverse Cardiac Events in Patients With Non-critical Coronary Artery Disease
Brief Title: Tissue-Type Plasminogen Activator (t-PA) Release Predicts Major Adverse Cardiac Events (MACE) in Patients With Non-critical Coronary Artery Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB# 030473; 5P5OHL081009-02 (Other: NIHLB)
Record Dates: First submitted 2009-03-19; First posted 2009-03-25 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Bradykinin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Bradykinin
  Interventions: Drug: Bradykinin

INTERVENTIONS:
Drug: Bradykinin — Bradykinin, 0.2 ug - 2ug/minute, one time intracoronary infusion over 6 minutes. Drug (bradykinin) will be infused into the left main coronary artery via diagnostic catheter (JL4) at an escalating rate of 0.2, 0.6, 2 g/ml (1ml/min). A 5F Multipurpose catheter will be advanced to coronary sinus for blood sampling.
  Other Names: Bachem Distribution Services GmbH-Bradykinin

SUMMARY:
Coronary artery disease is the leading cause of death in USA. Contemporary cardiac care has substantially reduced mortality and morbidity in patients with severe coronary artery disease. However, patients with mild to moderate coronary artery stenosis (<70% stenosis) often present in the future with life threatening acute coronary syndrome which carries significant mortality and morbidity. It is difficult to predict outcomes in these patients before the events because the lack of complete understanding of the mechanisms underlying acute coronary syndrome and the lack of reliable markers that will predict major adverse cardiac events (MACE). Tissue-type plasminogen activator (t-PA) is released from endothelial cells and a major factor that prevent thrombosis in the coronary artery, the cause of acute coronary syndrome. Endothelial dysfunction impairs t-PA release. Therefore, we hypothesize that patients with impaired coronary artery t-PA release will have significantly higher risk for future MACE due to intrinsic fibrinolytic dysfunction that leads to increased thrombosis risk.

To test this hypothesis, we will determine whether intrinsic endothelial fibrinolytic dysfunction predicts MACE in patients with non-significant CAD. The study will measure t-PA release mediated by bradykinin, a major mediator for t-PA release. This will involve infusion of bradykinin into left main coronary artery of individuals who have undergone routine cardiac catheterization (clinically indicated). We will take blood samples from the coronary sinus and measure t-PA and plasminogen activator inhibitor-1 antigen and activity levels.

DETAILED DESCRIPTION:
Tissue-type Plasminogen Activator (tPA) is a protein in the blood which breaks down clots and plays an important role in preventing myocardial infarction. It is produced by the endothelial cell lining of the blood vessels. Previous studies demonstrate that t-PA is released in response to the hormones bradykinin and acetylcholine. Impaired t-PA release upon bradykinin stimulation may indicate endothelial dysfunction that leads to the development of acute coronary syndrome. In this project, we will determine whether impaired t-PA release can predict future occurrence of acute coronary syndrome. The study will involve individuals getting routine left heart cardiac catheterizations (indication for cardiac catheterization is solely based on clinical indication). Prior to the procedure, patient will have two blood samples (5 ml each) collected from their forearm before and after 2 minutes blood pressure cuff inflation on their arm. After routine diagnostic cardiac catheterization and there is no severe coronary artery stenosis (<70% stenosis), research protocol will be initiated. Study includes infusion with increasing doses of bradykinin into their left main coronary artery, and sample small amounts of blood from their coronary sinus (15 ml total).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 year old male and female patients
2. All patients are referred for elective cardiac catheterization based on clinical indication
3. Cath shows mild or moderate (<70% stenosis) CAD that does not require mechanical intervention

Exclusion Criteria:

1. Severe stenosis requires intervention.
2. Significant left main coronary artery disease (>40%).
3. Acute MI or acute coronary syndrome with enzyme elevation or ischemic EKG changes
4. Patients with severe left ventricular dysfunction (EF<35%)
5. Prior history of myocardial infarction
6. History of stroke within 3 months.
7. Recent history of thrombolytic
8. History of coronary intervention within previous 6 months.
9. Patients with history of coronary spasm
10. Patients with congestive heart failure (class III and IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Vaughn, MD, Principal Investigator — Northwestern University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States